CLINICAL TRIAL: NCT02298361
Title: Innovative Methods for Parents And Clinics to Create Tools (IMPACCT) for Kids' Care
Brief Title: IMPACCT for Kids' Care
Acronym: IMPACCT
Status: Completed | Type: Observational
Sponsor: OCHIN, Inc. (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: PCORI Award (308)
Record Dates: First submitted 2014-11-05; First posted 2014-11-21 (Estimated); Results first posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-04

CONDITIONS: Insurance Status/Stability
Keywords: Adolescent; Child; Child Health Services/organization & administration*; Child, Preschool; Cohort Studies; Community Health Centers/organization & administration; Community Health Centers/standards; Electronic Health Records; Feasibility Studies; Female; Health Services Accessibility/economics; Humans; Infant; Infant, Newborn; Insurance Coverage; Insurance Coverage/statistics & numerical data; Insurance Coverage/trends; Insurance, Health; Insurance, Health/legislation & jurisprudence; Insurance, Health/statistics & numerical data; Insurance, Health/trends; Logistic Models; Longitudinal Studies; Male; Medicaid; Medicaid/statistics & numerical data; Medicaid/trends; Medicaid/utilization; Medically Uninsured; Medicare/statistics & numerical data; Medicare/trends; Medicare/utilization; Multivariate Analysis; Oregon; Patient Protection and Affordable Care Act; Patient-Centered Care; Pediatrics/legislation & jurisprudence; Pediatrics/standards; Population Surveillance/methods; Primary Health Care/economics; Quality Assurance, Health Care/legislation & jurisprudence; Quality Assurance, Health Care/methods; Quality Indicators, Health Care; Retrospective Studies; Socioeconomic Factors; United States; Young Adult
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Intervention patients: Community Health Centers that implemented health insurance outreach IT tools: active patients on whom tools were used
  Interventions: Other: Health insurance outreach IT tools
- Within-clinic comparison patients: Community Health Centers that implemented health insurance outreach IT tools: active patients on whom tools were not used
- Control clinic comparison patients: Matched Community Health Centers that did not implement health insurance outreach IT tools: active patients

INTERVENTIONS:
Other: Health insurance outreach IT tools — IT tools that support Community Health Centers in children's health insurance outreach efforts ("insurance outreach IT tools"), adapted from tools proven to support chronic disease management.
  Groups: Intervention patients

SUMMARY:
Health insurance is important for children. Public insurance programs are available to many children, but some families report being confused about how to get and keep this insurance. Community Health Centers (CHCs) can help families get and keep health insurance for their children.

The investigators will work with families, policy makers, and community health care providers and staff to develop and test new computer health information technology (IT) tools to help health care clinics find pediatric patients in need of insurance and communicate with their families about public insurance programs. These tools will be based on technologies currently used to help patients and clinics manage chronic diseases. The investigators will test the tools by comparing four clinics using the tools and four clinics not using the tools. The investigators will look to see if children in the clinics using the tools are more likely to have health insurance and also more likely to receive certain health care services, compared to children in the clinics without such tools. The investigators will also look at health insurance rates and health care services for a larger population of Oregon children.

DETAILED DESCRIPTION:
Summary of protocol changes made:

1. Changes to eligibility criteria. We changed patient eligibility to include all pediatric patients through age 19 with >=1 clinical visit in the study period. These decisions were based on: 1) at age 20, individuals are no longer eligible for children's Medicaid or CHIP in Oregon; 2) identification of PCP assignment was difficult in the EHR.
2. Added second comparison group/study arm. In the intervention clinics, the tools were used on a smaller number of pediatric patients than anticipated, and there were significant demographic differences between intervention and control site patients, despite the clinics being matched. Thus we added a second comparison group, "within-clinic comparison patients" as pediatric patients with >=1 visit at an intervention clinic in the study period but on whom the tools were NOT used. This provided a comparison group that accounted for clinic-level effects and was more demographically similar to the "intervention patients" on whom tools were used.
3. Revision of Aim 3 - CHIPRA recommended care assessment. We did not pursue assessment of CHIPRA quality care measures due to 1) limited follow-up time due to the need to implement iterative modifications to the study HIT tools, and 2) the tools were used on a smaller set of pediatric patients than anticipated, thus we had a very limited denominator for these analyses.

ELIGIBILITY:
Inclusion Criteria:

* age 0-19
* established patient (>=1 clinical visit at a study clinic in the assessment period)

Exclusion Criteria:

* age > 19
* not an established patient

Max Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: For the analysis of the primary study outcome, our study population will include all children who are "established" patients at an intervention or control clinic. Children will be considered "established" patients if they had >=1 clinical visit at a study clinic during the 18-month study period.
Sampling Method: Non-Probability Sample
Enrollment: 27251 (Actual)
Dates: Start 2013-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer DeVoe, MD, DPhil, Principal Investigator — OCHIN, OHSU; Christine Nelson, RN, PhD, Study Director — OCHIN, Inc.

REFERENCES:
- [Background] Devoe JE. Being uninsured is bad for your health: can medical homes play a role in treating the uninsurance ailment? Ann Fam Med. 2013 Sep-Oct;11(5):473-6. doi: 10.1370/afm.1541. PMID 24019280
- [Background] Angier H, Gold R, Crawford C, P O'Malley J, J Tillotson C, Marino M, DeVoe JE. Linkage methods for connecting children with parents in electronic health record and state public health insurance data. Matern Child Health J. 2014 Nov;18(9):2025-33. doi: 10.1007/s10995-014-1453-8. PMID 24562505
- [Background] DeVoe J, Angier H, Likumahuwa S, Hall J, Nelson C, Dickerson K, Keller S, Burdick T, Cohen D. Use of qualitative methods and user-centered design to develop customized health information technology tools within federally qualified health centers to keep children insured. J Ambul Care Manage. 2014 Apr-Jun;37(2):148-54. doi: 10.1097/JAC.0000000000000016. PMID 24594562
- [Background] DeVoe JE, Tillotson CJ, Angier H, Wallace LS. Predictors of children's health insurance coverage discontinuity in 1998 versus 2009: parental coverage continuity plays a major role. Matern Child Health J. 2015 Apr;19(4):889-96. doi: 10.1007/s10995-014-1590-0. PMID 25070735
- [Background] Hatch B, Angier H, Marino M, Heintzman J, Nelson C, Gold R, Vakarcs T, Devoe J. Using electronic health records to conduct children's health insurance surveillance. Pediatrics. 2013 Dec;132(6):e1584-91. doi: 10.1542/peds.2013-1470. Epub 2013 Nov 18. PMID 24249814
- [Background] Angier H, Likumahuwa S, Finnegan S, Vakarcs T, Nelson C, Bazemore A, Carrozza M, DeVoe JE. Using geographic information systems (GIS) to identify communities in need of health insurance outreach: An OCHIN practice-based research network (PBRN) report. J Am Board Fam Med. 2014 Nov-Dec;27(6):804-10. doi: 10.3122/jabfm.2014.06.140029. PMID 25381078
- [Background] DeVoe JE, Angier H, Burdick T, Gold R. Health information technology: an untapped resource to help keep patients insured. Ann Fam Med. 2014 Nov-Dec;12(6):568-72. doi: 10.1370/afm.1721. PMID 25384821
- [Background] Angier H, Hoopes M, Gold R, Bailey SR, Cottrell EK, Heintzman J, Marino M, DeVoe JE. An early look at rates of uninsured safety net clinic visits after the Affordable Care Act. Ann Fam Med. 2015 Jan-Feb;13(1):10-6. doi: 10.1370/afm.1741. PMID 25583886
- [Background] Heintzman J, Marino M, Hoopes M, Bailey SR, Gold R, O'Malley J, Angier H, Nelson C, Cottrell E, Devoe J. Supporting health insurance expansion: do electronic health records have valid insurance verification and enrollment data? J Am Med Inform Assoc. 2015 Jul;22(4):909-13. doi: 10.1093/jamia/ocv033. Epub 2015 Apr 17. PMID 25888586
- [Background] DeVoe JE, Crawford C, Angier H, O'Malley J, Gallia C, Marino M, Gold R. The Association Between Medicaid Coverage for Children and Parents Persists: 2002-2010. Matern Child Health J. 2015 Aug;19(8):1766-74. doi: 10.1007/s10995-015-1690-5. PMID 25874876
- [Background] Gold R, Burdick T, Angier H, Wallace L, Nelson C, Likumahuwa-Ackman S, Sumic A, DeVoe JE. Improve Synergy Between Health Information Exchange and Electronic Health Records to Increase Rates of Continuously Insured Patients. EGEMS (Wash DC). 2015 Aug 6;3(1):1158. doi: 10.13063/2327-9214.1158. eCollection 2015. PMID 26355818
- [Background] DeVoe JE, Tillotson CJ, Marino M, O'Malley J, Angier H, Wallace LS, Gold R. Trends in Type of Health Insurance Coverage for US Children and Their Parents, 1998-2011. Acad Pediatr. 2016 Mar;16(2):192-9. doi: 10.1016/j.acap.2015.06.009. Epub 2015 Aug 18. PMID 26297668
- [Background] Angier H, Marino M, Sumic A, O'Malley J, Likumahuwa-Ackman S, Hoopes M, Nelson C, Gold R, Cohen D, Dickerson K, DeVoe JE. Innovative methods for parents and clinics to create tools for kids' care (IMPACCT Kids' Care) study protocol. Contemp Clin Trials. 2015 Sep;44:159-163. doi: 10.1016/j.cct.2015.08.010. Epub 2015 Aug 18. PMID 26291916
- [Background] Arkind J, Likumahuwa-Ackman S, Warren N, Dickerson K, Robbins L, Norman K, DeVoe JE. Lessons Learned from Developing a Patient Engagement Panel: An OCHIN Report. J Am Board Fam Med. 2015 Sep-Oct;28(5):632-8. doi: 10.3122/jabfm.2015.05.150009. PMID 26355135
- [Background] Likumahuwa-Ackman S, Angier H, Sumic A, Harding RL, Cottrell EK, Cohen DJ, Nelson CA, Burdick TE, Wallace LS, Gallia C, DeVoe JE. IMPACCT Kids' Care: a real-world example of stakeholder involvement in comparative effectiveness research. J Comp Eff Res. 2015 Aug;4(4):351-7. doi: 10.2217/cer.15.24. PMID 26274796
- [Background] Hoopes MJ, Angier H, Gold R, Bailey SR, Huguet N, Marino M, DeVoe JE. Utilization of Community Health Centers in Medicaid Expansion and Nonexpansion States, 2013-2014. J Ambul Care Manage. 2016 Oct-Dec;39(4):290-8. doi: 10.1097/JAC.0000000000000123. PMID 26765808
- [Background] Hatch B, Tillotson C, Angier H, Marino M, Hoopes M, Huguet N, DeVoe J. Using the electronic health record for assessment of health insurance in community health centers. J Am Med Inform Assoc. 2016 Sep;23(5):984-90. doi: 10.1093/jamia/ocv179. Epub 2016 Jan 23. PMID 26911812
- [Derived] DeVoe JE, Hoopes M, Nelson CA, Cohen DJ, Sumic A, Hall J, Angier H, Marino M, O'Malley JP, Gold R. Electronic health record tools to assist with children's insurance coverage: a mixed methods study. BMC Health Serv Res. 2018 May 10;18(1):354. doi: 10.1186/s12913-018-3159-x. PMID 29747644

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Patients | Within-clinic Comparison Patients | Control Clinic Comparison Patients
Started | 2240 | 12784 | 12227
Completed | 2240 | 12784 | 12227
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Patients | Within-clinic Comparison Patients | Control Clinic Comparison Patients | Total
Number analyzed (Participants) | 2240 | 12784 | 12227 | 27251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2170 | 12306 | 11783 | 26259
  Between 18 and 65 years | 70 | 478 | 444 | 992
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (5.4) | 8.6 (5.9) | 8.2 (5.9) | 8.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1119 | 6524 | 6128 | 13771
  Male | 1121 | 6260 | 6099 | 13480
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2128 | 8270 | 7266 | 17664
  Not Hispanic or Latino | 103 | 4031 | 4831 | 8965
  Unknown or Not Reported | 9 | 483 | 130 | 622
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 26 | 166 | 194
  Asian | 8 | 198 | 297 | 503
  Native Hawaiian or Other Pacific Islander | 3 | 30 | 128 | 161
  Black or African American | 17 | 407 | 1345 | 1769
  White | 1996 | 10758 | 8462 | 21216
  More than one race | 1 | 26 | 260 | 287
  Unknown or Not Reported | 213 | 1339 | 1569 | 3121
Primary language [Number; unit: participants]
  Spanish | 1976 | 6490 | 5803 | 14269
  English | 241 | 5629 | 5103 | 10973
  Other | 22 | 622 | 1125 | 1769
  Unknown | 1 | 43 | 196 | 240
Household income as percent of Federal Poverty Level [Number; unit: participants]
  <=138% FPL | 2083 | 11253 | 9998 | 23334
  139-199% FPL | 114 | 734 | 918 | 1766
  >=200% FPL | 29 | 283 | 1204 | 1516
  Unknown | 14 | 514 | 107 | 635

OUTCOME MEASURES:

1. Primary Outcome: Percent of Study Period Covered by Medicaid
Description: Percent of total days in 22-month assessment period that each child was covered by Medicaid insurance. Assessed using state administrative records linked to EHR data; this outcome was assessed among the subset of participants with a Medicaid ID (and thus could be linked between the two data sources).
Time Frame: 6 months pre- through 16 months post-tool implementation
Measure: Number; unit: participants
Arm/Group | Intervention Patients | Within-clinic Comparison Patients | Control Clinic Comparison Patients
Number analyzed (Participants) | 2080 | 11534 | 11729
participants
  0% covered | 30 | 451 | 297
  1-49% covered | 113 | 1062 | 933
  50-99% covered | 648 | 3198 | 3386
  100% covered | 1289 | 6823 | 7113

2. Primary Outcome: Proportion of Patients Who Gained Medicaid Coverage
Description: Proportion of participants who gained Medicaid coverage after a period of uninsurance. Assessed using state administrative records linked to EHR data; this outcome was assessed among the subset of participants with a Medicaid ID (and thus could be linked between the two data sources) and who had partial coverage during the study period (i.e., patients with 100% coverage were not 'eligible' to gain coverage).
Time Frame: 6 months pre- through 16 months post-tool implementation
Measure: Number; unit: participants
Arm/Group | Intervention Patients | Within-clinic Comparison Patients | Control Clinic Comparison Patients
Number analyzed (Participants) | 761 | 4260 | 4319
participants | 444 | 2611 | 2426
Statistical Analysis 1: Comparison: Intervention Patients vs Within-clinic Comparison Patients; Test type: Superiority or Other; Generalized estimating equation; GEE model clustered by clinic, adjusted for demographics, number of visits, new/established patient at first visit, and household factors; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.60 to 1.93] — Adjusted odds of gaining Medicaid: intervention patients (numerator) relative to within-clinic comparison patients (denominator)
Statistical Analysis 2: Comparison: Intervention Patients vs Control Clinic Comparison Patients; Test type: Superiority or Other; Generalized estimating equation; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.28, 95% CI 2-sided [1.91 to 2.72] — Adjusted odds of gaining Medicaid: intervention patients (numerator) relative to control clinic comparison patients (denominator)

3. Primary Outcome: Proportion of Patients Who Lost Medicaid Coverage
Description: Proportion of participants who lost Medicaid coverage after a period of insurance. Assessed using state administrative records linked to EHR data; this outcome was assessed among the subset of participants with a Medicaid ID (and thus could be linked between the two data sources) and who had partial coverage during the study period (i.e., patients with 100% coverage were not 'eligible' to lose coverage).
Time Frame: 6 months pre- through 16 months post-tool implementation
Measure: Number; unit: participants
Arm/Group | Intervention Patients | Within-clinic Comparison Patients | Control Clinic Comparison Patients
Number analyzed (Participants) | 761 | 4260 | 4319
participants | 377 | 1873 | 2173
Statistical Analysis 1: Comparison: Intervention Patients vs Within-clinic Comparison Patients; Test type: Superiority or Other; Generalized estimating equation; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.53 to 0.94] — Adjusted odds of losing Medicaid: intervention patients (numerator) relative to within-clinic comparison patients (denominator)
Statistical Analysis 2: Comparison: Intervention Patients vs Control Clinic Comparison Patients; Test type: Superiority or Other; Generalized estimating equation; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.45 to 0.67] — Adjusted odds of losing Medicaid: intervention patients (numerator) relative to control clinic comparison patients (denominator)

ADVERSE EVENTS:
Description: Adverse events not monitored; not applicable to the study.
Arm/Group | Intervention Patients | Within-clinic Comparison Patients | Control Clinic Comparison Patients
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No